CLINICAL TRIAL: NCT04603625
Title: Postural Management to Prevent Hip Luxation in Quadriplegic Cerebral Palsy Children: Comparing Two Approaches in a Randomized Controlled Trial
Brief Title: Postural Management for Hip Luxation in Quadriplegic Cerebral Palsy
Acronym: CPluxprev2020
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Ospedale IRCCS G. Gaslini di Genova (Unknown); IRCCS Eugenio Medea (Other); IRCCS Don Carlo Gnocchi di Firenze (Unknown); Azienda Unita' Sanitaria Locale Di Modena (Other); Azienda Usl di Bologna (Other Government); Azienda Unità Sanitaria Locale della Romagna (Other); Azienda ULSS di Verona e Provincia (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 723/2020/SPER/AUSLRE
Record Dates: First submitted 2020-10-01; First posted 2020-10-27 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-02

CONDITIONS: Quadriplegic Cerebral Palsy
Keywords: hip luxation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Physicians measuring Migration Percentage (Primary Outcome) will be blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sitting position centering femoral heads (Experimental): sitting position centering femoral heads according to Lespargot diagram
  Interventions: Other: postural management
- Usual postural management (Active Comparator): sitting with the trunk aligned and hips abducted to facilitate activities of daily living
  Interventions: Other: postural management

INTERVENTIONS:
Other: postural management — postural management in sitting position

SUMMARY:
Cerebral palsy (CP) is the most common motor disability in childhood. Among these, hip luxation represents the most frequent and clinically relevant one, affecting 72% of non-ambulatory CP children. Reconstructive surgical treatment is debated in severe CP children, for whom it is crucial to identify an effective preventive approach. The aim of our study is to verify if keeping a sitting position centering femoral heads is more effective than usual postural management (sitting with the trunk aligned and hips abducted), in preventing hip luxation in quadriplegic CP children. It's a multicenter randomized controlled study (13 sites involved). A total of 102 quadriplegic CP children, aged 1-6 years-old, classified as Gross Motor Function Measure System 4 or 5, will be recruited and randomized to usual or experimental sitting, at least 5 hours a day, for 2 years. The primary outcome will be the degree of luxation, measured by means of the Migration Percentage (MP), on pelvic radiography, at 12 and 24 months. Secondary outcomes will include compliance and Health Related-Quality of Life, using validated tools, hip pain, device cost, MRI lesions, concurrent direct neuromotor treatment, use of standing devices and spasticity treatments (botulinum toxin, per os or intrathecal baclofen, selective dorsal rhizotomy). Experimental sitting is expected to reduce the MP change compared to usual care. It will be of interest to compare compliance, QoL and costs in either groups: aspects affecting the effectiveness. Furthermore to evaluate correlations between MP and spasticity treatments, MRI lesion type, and other clinical features.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy spastic or dyskinetic
* GMFCS 4 or 5
* MP<41%
* Informed Consent acquired

Exclusion Criteria:

* muscle contracture overcoming defined passive Range Of Motion (ROM)limits
* anterior hip luxation
* previous reconstructive hip surgery
* preventive surgery in previous 12 months
* lumbar scoliosis >20° Cobb

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Migration Percentage | Day 0, Month 12, Months 24
  measure of hip luxation on pelvic radiography

SECONDARY OUTCOMES:
Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) | Day 0, Month 12, Month 24
  Parents will fill in a questionnaire about Health Related Quality of Life referred to their child. Minimum value 0, maximum value 100, higher scores mean a better outcome.
Quebec User Evaluation of Satisfaction with Assistive Technology (IT-QUEST) | Month 12, Month 24
  Parents will fill in a questionnaire measuring their satisfaction about the assistive device ensuring the desired sitting position of their child. Minimum value 1, maximum value 5,higher scores mean a better outcome.
Incidence of pain | Day 0, Month 6, Month 12, Month 18, Month 24
  Care givers will be interviewed about presence or absence of hip pain in the previous months during personal care and activities of daily living
Assistive devices costs | Day 0, Month 6, Month 12, Month 18, Month 24
  Costs paid by Health Institution for sitting systems used during the study
Percentage of patients attending Botulinum Toxin-A injections | Day 0, Month 6, Month 12, Month 18, Month 24
  Botulinum Toxin-A injections in muscles around the hip during the study will be recorded
Percentage of patients attending direct physical treatment | Day 0, Month 6, Month 12, Month 18, Month 24
  Physiotherapy, other Neuromotor Therapy during the study
Percentage of patients using standing devices in abduction | Day 0, Month 6, Month 12, Month 18, Month 24
  It will be recorded if the patients will be using standing devices at least 5 hours/week, less than 5 h/week or never
Type of CP (Dyskinetic or spastic) | Day 0
  Type of CP will be recorded to evaluate any association with MP change
Percentage of patients having Intrathecal Baclofen (ITB) | Day 0
  It will be recorded if patients have ITB to evaluate any association with MP change
Percentage of patients taking Baclofen per os | Day 0, Month 6, Month 12, Month 18, Month 24
  Baclofen oral medication during the study will be recorded
Percentage of patients who underwent Selective Dorsal Rhizotomy (SDR) | Day 0
  It will be recorded if patients underwent SDR in the past to evaluate any association with MP change
Age | Day 0
  Age will be recorded to evaluate any association with MP change
Sex | Day 0
  Sex will be recorded to evaluate any association with MP change
Type of lesion at MRI | Day 0
  Type of lesion at MRI, according to Neonatal Neuroimaging Classification System (maldevelopments | predominant white matter injury | predominant grey matter injury | miscellaneous | Normal). Data will be registered based on previously acquired MRI, considering that the exam is mandatory for the diagnosis of cerebral palsy. It will be recorded to evaluate any association with MP change

CONTACTS AND LOCATIONS:
Overall Officials: SILVIA FACCIOLI, Study Chair — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Azienda Unità Sanitaria Locale Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No
We are going to share results and data at the end of the study by publication

REFERENCES:
- [Background] Bouwhuis CB, van der Heijden-Maessen HC, Boldingh EJ, Bos CF, Lankhorst GJ. Effectiveness of preventive and corrective surgical intervention on hip disorders in severe cerebral palsy: a systematic review. Disabil Rehabil. 2015;37(2):97-105. doi: 10.3109/09638288.2014.908961. Epub 2014 Apr 14. PMID 24731007
- [Background] Dalen Y, Saaf M, Ringertz H, Klefbeck B, Mattsson E, Haglund-Akerlind Y. Effects of standing on bone density and hip dislocation in children with severe cerebral palsy. Adv Physiother,2010;12:187-93.
- [Background] Diab M, Staheli LT. Ortopedia Pediatrica, 3° ed., Verduci ed., p.65
- [Background] Galeoto G, Colucci M, Guarino D, Esposito G, Cosma E, De Santis R, Grifoni G, Valente D, Tofani M. Exploring Validity, Reliability, and Factor Analysis of the Quebec User Evaluation of Satisfaction with Assistive Technology in an Italian Population: A Cross-Sectional Study. Occup Ther Health Care. 2018 Oct;32(4):380-392. doi: 10.1080/07380577.2018.1522682. Epub 2018 Dec 31. PMID 30596451
- [Background] Hagglund G, Goldring M, Hermanson M, Rodby-Bousquet E. Pelvic obliquity and measurement of hip displacement in children with cerebral palsy. Acta Orthop. 2018 Dec;89(6):652-655. doi: 10.1080/17453674.2018.1519104. Epub 2018 Oct 17. PMID 30326758
- [Background] Hagglund G, Lauge-Pedersen H, Wagner P. Characteristics of children with hip displacement in cerebral palsy. BMC Musculoskelet Disord. 2007 Oct 26;8:101. doi: 10.1186/1471-2474-8-101. PMID 17963501
- [Background] • Lespargot A. La luxation postéro-externe de la hanche chez l'enfant IMC ou polyhandicapé. Motricité cérébrale,1991;12:37-61
- [Background] Lins LAB, Watkins CJ, Shore BJ. Natural History of Spastic Hip Disease. J Pediatr Orthop. 2019 Jul;39(Issue 6, Supplement 1 Suppl 1):S33-S37. doi: 10.1097/BPO.0000000000001347. PMID 31169645
- [Background] Martinsson C, Himmelmann K. Effect of weight-bearing in abduction and extension on hip stability in children with cerebral palsy. Pediatr Phys Ther. 2011 Summer;23(2):150-7. doi: 10.1097/PEP.0b013e318218efc3. PMID 21552077
- [Background] Gmelig Meyling C, Ketelaar M, Kuijper MA, Voorman J, Buizer AI. Effects of Postural Management on Hip Migration in Children With Cerebral Palsy: A Systematic Review. Pediatr Phys Ther. 2018 Apr;30(2):82-91. doi: 10.1097/PEP.0000000000000488. PMID 29578990
- [Background] Miller SD, Juricic M, Hesketh K, Mclean L, Magnuson S, Gasior S, Schaeffer E, O'donnell M, Mulpuri K. Prevention of hip displacement in children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2017 Nov;59(11):1130-1138. doi: 10.1111/dmcn.13480. Epub 2017 Jun 2. PMID 28574172
- [Background] Narayanan UG, Fehlings D, Weir S, Knights S, Kiran S, Campbell K. Initial development and validation of the Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD). Dev Med Child Neurol. 2006 Oct;48(10):804-12. doi: 10.1017/S0012162206001745. PMID 16978459
- [Background] Picciolini O, LE Metayer M, Consonni D, Cozzaglio M, Porro M, Gasparroni V, Panou A, Mosca F, Portinaro NM. Can we prevent hip dislocation in children with cerebral palsy? Effects of postural management. Eur J Phys Rehabil Med. 2016 Oct;52(5):682-690. Epub 2016 May 6. PMID 27153480
- [Background] Sproccati N, Bertana S, Battisti N, Feliciangeli A, Baroncini C, Zenesini C, Cersosimo A. Italian translation and cross-cultural adaptation of the questionnaire for the assessment of quality of life in children with cerebral palsy: Caregiver priorities and Child Health Index of Life with disabilities. Minerva Med. 2021 Oct;112(5):651-653. doi: 10.23736/S0026-4806.19.06072-5. Epub 2019 Jun 25. No abstract available. PMID 31256575
- [Background] Terjesen T. The natural history of hip development in cerebral palsy. Dev Med Child Neurol. 2012 Oct;54(10):951-7. doi: 10.1111/j.1469-8749.2012.04385.x. Epub 2012 Aug 13. PMID 22881288
- [Background] Wynter M, Gibson N, Willoughby KL, Love S, Kentish M, Thomason P, Graham HK; National Hip Surveillance Working Group. Australian hip surveillance guidelines for children with cerebral palsy: 5-year review. Dev Med Child Neurol. 2015 Sep;57(9):808-20. doi: 10.1111/dmcn.12754. Epub 2015 Apr 3. PMID 25846730
- [Derived] Faccioli S, Maggi I, Pagliano E, Migliorini C, Michelutti A, Guerra L, Ronchetti A, Cristella G, Battisti N, Mancini L, Picciolini O, Alboresi S, Trabacca A, Kaleci S. Sitting Postural Management to Prevent Migration Percentage Progression in Non-Ambulatory Children with Cerebral Palsy: Randomized Controlled Trial Preliminary Data. J Clin Med. 2024 May 27;13(11):3129. doi: 10.3390/jcm13113129. PMID 38892841